CLINICAL TRIAL: NCT04377997
Title: A Randomized, Open-Label Trial of Therapeutic Anticoagulation in COVID-19 Patients With an Elevated D-Dimer
Brief Title: Safety and Efficacy of Therapeutic Anticoagulation on Clinical Outcomes in Hospitalized Patients With COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rahul Sakhuja, M.D., Interventional Cardiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020P001136
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Diseases; COVID-19
MeSH Terms: conditions — Cardiovascular Diseases; COVID-19 | interventions — Enoxaparin; Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Therapeutic Anticoagulation Group (Experimental): Patients identified as eligible through discussions with the primary care team and review of the electronic medical record will be approached and consented as described above in "Subject Enrollment" and "Procedures for obtaining consent".
  For research purposes, 20ml of blood will be drawn and stored for biobanking at the following timepoints: at baseline (i.e., after enrollment and before randomization), 5-7 days post-randomization, and on the day of discharge. The blood sample taken at baseline will also be used to conduct a pregnancy test for women of childbearing age.
  After enrollment and blood collection, patients will then be randomized to therapeutic anticoagulation (LMWH for most subjects but UFH for those with morbid obesity or moderate to severe renal dysfunction as noted below) or standard of care anticoagulation. Those assigned to the therapeutic anticoagulation group will receive a higher dose of heparin.
  Interventions: Drug: Enoxaparin
- Standard of Care Anticoagulation Group (Active Comparator): Patients identified as eligible through discussions with the primary care team and review of the electronic medical record will be approached and consented as described above in "Subject Enrollment" and "Procedures for obtaining consent".
  For research purposes, 20ml of blood will be drawn and stored for biobanking at the following timepoints: at baseline (i.e., after enrollment and before randomization), 5-7 days post-randomization, and on the day of discharge. The blood sample taken at baseline will also be used to conduct a pregnancy test for women of childbearing age.
  After enrollment and blood collection, patients will then be randomized to therapeutic anticoagulation or standard of care anticoagulation. Those assigned to the standard of care anticoagulation group will receive the normal dose of heparin as per the Mass General guidelines.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Given the established link between endothelial dysfunction and thrombosis in patients with cardiovascular disease9, 10 and the association between coagulopathy and adverse outcomes in patients with sepsis11, the association between increased coagulation activity, end-organ injury, and mortality risk may represent a modifiable risk factor among COVID-19 patients with critical illness. Therefore, we propose to conduct a randomized, open-label trial of therapeutic anticoagulation in COVID-19 patients with an elevated D-dimer to evaluate the efficacy. Most patients will receive low molecular weight heparin however, unfractionated heparin (UFH) will be administered for those with morbid obesity or moderate to severe renal dysfunction.
  Other Names: Heparin; Low molecular weight heparin

SUMMARY:
The coronavirus disease 2019 (COVID-19) global pandemic caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has caused considerable morbidity and mortality in over 170 countries. Increasing age and burden of cardiovascular comorbidities are associated with a worse prognosis among patients with COVID-19. In addition, serologic markers of more severe disease including coagulation abnormalities and thrombocytopenia, are not uncommon among patients hospitalized with severe COVID-19 infection and are more common in patients who died in-hospital. As the COVID-19 pandemic continues to grow, there is a pressing need to identify safe, effective, and widely available therapies that can be scaled and rapidly incorporated into clinical practice. Understanding the putative mechanism of increased mortality risk associated with abnormal coagulation function and cardiac injury is critical to guide studies of promising therapeutic interventions. Published and anecdotal reports indicate that endothelial dysfunction and thrombosis are common in critically ill patients with COVID-19, including reports of diffuse microvascular thrombosis in the lungs, heart, liver, and kidneys. Patients with cardiovascular disease (CVD) and CVD risk factors are known to have endothelial dysfunction and a heightened risk of thrombosis. A recent study of COVID-19 inpatients from Wuhan, China observed that an elevated D-dimer level greater than 1 ug/mL was associated with an 18 times higher risk of in-hospital death, underscoring the importance of increased coagulation activity as a potential modifiable risk marker that may drive end-organ injury. Given the established link between endothelial dysfunction and thrombosis in patients with cardiovascular disease, and the association between coagulopathy and adverse outcomes in patients with sepsis, the association between increased coagulation activity, end-organ injury, and mortality risk may represent a modifiable risk factor among COVID-19 patients with critical illness. Therefore, we propose to conduct a randomized, open-label trial of therapeutic anticoagulation in COVID-19 patients with an elevated D-dimer to evaluate the efficacy and safety.

DETAILED DESCRIPTION:
Patients identified as eligible through discussions with the primary care team and review of the electronic medical record will be approached and consented as described above in "Subject Enrollment" and "Procedures for obtaining consent".

For research purposes, 20mL of blood will be drawn and stored for biobanking at the following timepoints: at baseline (i.e., after enrollment and before randomization), 5-7 days post-randomization, and on the day of discharge.

After enrollment and blood collection, patients will then be randomized to therapeutic anticoagulation (LMWH for most subjects but UFH for those with morbid obesity or moderate to severe renal dysfunction as noted below) or standard of care.

Based on the MGH COVID-19 Treatment Guidance document, the risk stratification recommends daily complete blood count (CBC), comprehensive metabolic panel (CMP), creatine kinase (CPK), ferritin, C-reactive protein (CRP), and erythrocyte sedimentation rate (ESR). In addition, PT, PTT, fibrinogen, and D-dimer are recommended to be checked every other day if in the ICU or daily if elevated. Given that by virtue of the inclusion criteria of our study (i.e., a D-dimer >1ug/mL), all of our patients will be within Category 3 and all of the above markers will be obtained for clinical purposes and thus will also be documented for research purposes. For clinical risk stratification, LDH is to be checked daily if elevated and troponin to be checked q2-3d if elevated. If clinically indicated, procalcitonin will be measured and IL-6 obtained in patients in Category 2 or 3 disease severity. If measured for clinical purposes, LDH, troponin, procalcitonin, and IL-6 will be recorded for research purposes.

ELIGIBILITY:
Inclusion:

* COVID-19 positive on admission or during hospitalization (having been tested within the past 5 days) with symptoms consistent with COVID-19 including fever (≥ 38C, 100.4F), pneumonia, symptoms of lower respiratory illness (e.g., cough, difficulty breathing), loss of smell or taste, myalgias, pharyngitis, or diarrhea
* Admitted to the regular medical floor or intensive care unit (ICU) without severe ARDS (P/F ratio<100)
* Elevated D-dimer (>1.5g/mL)
* Age>18 years and not older than 90
* Fibrinogen >100
* Platelets >50,000
* No prior intracranial hemorrhage or recent ischemic stroke or TIA within 6 months
* D-dimer > 1500 ng/ml
* No other clinical indication for therapeutic anticoagulation (e.g., deep vein thrombosis [DVT], pulmonary embolism [PE], atrial fibrillation, acute coronary syndromes, or extracorporeal membrane oxygenation)

Exclusion:

* Disseminated intravascular coagulation (DIC) according to the International Society on Thrombosis and Hemostasis overt DIC definition
* Hemoglobin (Hgb) <8 g/dl
* Hypersensitivity to heparin or heparin formulation including heparin-induced thrombocytopenia
* Thrombocytopenia: platelets<50,000 platelets/ul
* Uncontrolled or active/recent bleeding including intracranial hemorrhage, signs of active bleeding (e.g., blood transfusion within 30 days), any GI bleed within the past 6 months, or internal bleeding within the past 1 month
* High bleeding risk: significant closed-head or facial trauma within 3 months, traumatic or prolonged CPR (>10min), or use of dual anti-platelet therapy
* Known or suspected pregnancy
* Recent (<48 hours) or planned spinal or epidural anesthesia or puncture
* If the patient is on other anticoagulants, antihistamines, nonsteroidal anti-inflammatory drugs (i.e. aspirin) or hydroxychloroquine
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with the composite efficacy endpoint of death, cardiac arrest, symptomatic deep venous thrombosis, pulmonary embolism, arterial thromboembolism, myocardial infarction, or hemodynamic shock. | 12 weeks
  Aim 1 - Risk of death, cardiac arrest, symptomatic deep venous thrombosis, pulmonary embolism, arterial thromboembolism, myocardial infarction, or hemodynamic shock.
Number of patients with a major bleeding event according to the International Society on Thrombosis and Haemostasis (ISTH) definition. | 12 weeks
  Aim 2 - Risk of major bleeding event according to the International Society on Thrombosis and Haemostasis (ISTH) definition.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Sakhuja, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Abdurahman Khalil, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] The Novel Coronavirus Pneumonia Emergency Response Epidemiology Team. The Epidemiological Characteristics of an Outbreak of 2019 Novel Coronavirus Diseases (COVID-19) - China, 2020. China CDC Wkly. 2020 Feb 21;2(8):113-122. No abstract available. PMID 34594836
- [Background] Schindler TH, Dilsizian V. Coronary Microvascular Dysfunction: Clinical Considerations and Noninvasive Diagnosis. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 1):140-155. doi: 10.1016/j.jcmg.2018.11.036. Epub 2019 Apr 12. PMID 30982670
- [Background] Dellinger RP. Inflammation and coagulation: implications for the septic patient. Clin Infect Dis. 2003 May 15;36(10):1259-65. doi: 10.1086/374835. Epub 2003 May 8. PMID 12746771
- [Background] Young E. The anti-inflammatory effects of heparin and related compounds. Thromb Res. 2008;122(6):743-52. doi: 10.1016/j.thromres.2006.10.026. Epub 2007 Aug 28. PMID 17727922
- [Result] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Frencken JF, Donker DW, Spitoni C, Koster-Brouwer ME, Soliman IW, Ong DSY, Horn J, van der Poll T, van Klei WA, Bonten MJM, Cremer OL. Myocardial Injury in Patients With Sepsis and Its Association With Long-Term Outcome. Circ Cardiovasc Qual Outcomes. 2018 Feb;11(2):e004040. doi: 10.1161/CIRCOUTCOMES.117.004040. PMID 29378734
- [Result] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Result] C. P. COVID-19: Abnormal Clotting Common in More Severe Disease. 2020.
- [Result] Chan MY, Andreotti F, Becker RC. Hypercoagulable states in cardiovascular disease. Circulation. 2008 Nov 25;118(22):2286-97. doi: 10.1161/CIRCULATIONAHA.108.778837. No abstract available. PMID 19029477
- [Result] Zarychanski R, Doucette S, Fergusson D, Roberts D, Houston DS, Sharma S, Gulati H, Kumar A. Early intravenous unfractionated heparin and mortality in septic shock. Crit Care Med. 2008 Nov;36(11):2973-9. doi: 10.1097/CCM.0b013e31818b8c6b. PMID 18824906
- [Result] Jaimes F, De La Rosa G, Morales C, Fortich F, Arango C, Aguirre D, Munoz A. Unfractioned heparin for treatment of sepsis: A randomized clinical trial (The HETRASE Study). Crit Care Med. 2009 Apr;37(4):1185-96. doi: 10.1097/CCM.0b013e31819c06bc. PMID 19242322
- [Result] Safety of Heparin in Patients with Septic Shock.
- [Result] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Result] Iba T, Levy JH, Warkentin TE, Thachil J, van der Poll T, Levi M; Scientific and Standardization Committee on DIC, and the Scientific and Standardization Committee on Perioperative and Critical Care of the International Society on Thrombosis and Haemostasis. Diagnosis and management of sepsis-induced coagulopathy and disseminated intravascular coagulation. J Thromb Haemost. 2019 Nov;17(11):1989-1994. doi: 10.1111/jth.14578. Epub 2019 Aug 13. No abstract available. PMID 31410983
- [Result] Zarychanski R, Abou-Setta AM, Kanji S, Turgeon AF, Kumar A, Houston DS, Rimmer E, Houston BL, McIntyre L, Fox-Robichaud AE, Hebert P, Cook DJ, Fergusson DA; Canadian Critical Care Trials Group. The efficacy and safety of heparin in patients with sepsis: a systematic review and metaanalysis. Crit Care Med. 2015 Mar;43(3):511-8. doi: 10.1097/CCM.0000000000000763. PMID 25493972
- [Result] Zidane M, Schram MT, Planken EW, Molendijk WH, Rosendaal FR, van der Meer FJ, Huisman MV. Frequency of major hemorrhage in patients treated with unfractionated intravenous heparin for deep venous thrombosis or pulmonary embolism: a study in routine clinical practice. Arch Intern Med. 2000 Aug 14-28;160(15):2369-73. doi: 10.1001/archinte.160.15.2369. PMID 10927736
- [Result] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Result] Morris TA, Castrejon S, Devendra G, Gamst AC. No difference in risk for thrombocytopenia during treatment of pulmonary embolism and deep venous thrombosis with either low-molecular-weight heparin or unfractionated heparin: a metaanalysis. Chest. 2007 Oct;132(4):1131-9. doi: 10.1378/chest.06-2518. Epub 2007 Jul 23. PMID 17646239
- [Result] Stein PD, Hull RD, Matta F, Yaekoub AY, Liang J. Incidence of thrombocytopenia in hospitalized patients with venous thromboembolism. Am J Med. 2009 Oct;122(10):919-30. doi: 10.1016/j.amjmed.2009.03.026. Epub 2009 Aug 13. PMID 19682670